CLINICAL TRIAL: NCT06877247
Title: A Mass Balance Study of [14C] SHR6508 in Chinese Hemodialysis Subjects With Secondary Hyperparathyroidism
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR6508-103
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] SHR6508 Injection Group (Experimental)
  Interventions: Drug: [14C] SHR6508 Injection

INTERVENTIONS:
Drug: [14C] SHR6508 Injection — [14C] SHR6508 injection.

SUMMARY:
The study is being conducted to determine the mass balance and routes of excretion of total radioactivity after the dose of [14C] SHR6508.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide a written informed consent form.
2. Male subjects and postmenopausal women.
3. Meet the Body Mass Index (BMI) standard.

Exclusion Criteria:

1. Subjects with a history of cardiovascular diseases.
2. Subjects with gastrointestinal diseases.
3. Subjects with a history of surgery.
4. Subjects with a history of blood loss.
5. Abnormal blood pressure.
6. Be allergic to a drug ingredient or component.
7. Subject with a history of alcohol abuse and drug abuse
8. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative excretion of radioactivity | Day 1 to Day 168.
Percentage of parent drug and its metabolites in plasma as a percentage of total radioactive exposure (%AUC) | Day 1 to Day 6.

SECONDARY OUTCOMES:
Adverse Events (AEs) | About 24 weeks.
Serious adverse Events (SAEs) | About 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided